CLINICAL TRIAL: NCT05794009
Title: An E-therapist: an Interactive Immersive Virtual Reality Exercise Program for People with Type 2 Diabetes
Brief Title: Virtual Reality Exercise Program for People with Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr YU Clare Chung Wah, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0036522
Record Dates: First submitted 2023-03-06; First posted 2023-03-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-03

CONDITIONS: Exercise Therapy
Keywords: exercise, diabetes, cognitive function, virtual reality
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Recruited participants from community centers will be randomly allocated into either an IVRE program or a home-based exercise program that is identical to the intervention group (control group) using computer-generated random numbers. This will be a single-blinded randomized controlled trial (RCT), where outcome assessor(s) will be blinded to the allocation of participants throughout the study. Participants will be informed of their allocated exercise protocols, and they will be advised not to disclose their allocated intervention to the assessor(s) or other participants.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor(s) will be blinded to the allocation of participants throughout the study. The name of the participants and the allocation will be removed from the assessment sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immersive Virtual Reality Exercise (IVRE) (Experimental): VR exercise training for at least three times a week for 12 consecutive weeks (a total of 36 sessions) guided by the e-therapist: The tailored VR-based exercise program involves aerobic and resistance exercises, and VR games.
  Interventions: Other: Immersive Virtual Reality Exercise (IVRE)
- Home Exercise (Active Comparator): Individuals randomized to the control group will attend a briefing session prior to the start of the program to complete demographic data collection and physical assessment. They will be given an exercise booklet and guided through a set of home-based exercises (identical training to the intervention group except for VR games) in the briefing session. Stepping exercises will be implemented as a substitution of cycling as an aerobic exercise training at home.
  Interventions: Other: Home Exercise

INTERVENTIONS:
Other: Immersive Virtual Reality Exercise (IVRE) — The IVRE program will include aerobic exercise, muscle strengthening exercise, balance and flexibility exercise.
  Arms: Immersive Virtual Reality Exercise (IVRE)
Other: Home Exercise — Aerobic exercise, muscle strengthening exercise, balance and flexibility exercise at home.
  Arms: Home Exercise

SUMMARY:
The purpose of this study is to examine the effectiveness of a virtual reality (VR) based rehabilitation protocol for improvement of blood glucose control and exercise compliance of patients.

Subjects aged 55-85 diagnosed with Type 2 diabetes will be recruited. A written consent will be obtained from subjects. Subjects recruited will be randomly divided into one of the two groups. The VR group will receive an exercise program conducted in elderly centre or a control group will receive home exercise program. The 12-week exercise program will be conducted three times per week and each session will last for one hour. Assessment that takes about one hour to complete will be carried out at baseline, mid-way (6th week) and after the 12-week exercise training. Assessment items include physical, psychosocial and cognitive function. Also, blood test on HbA1c will be carried out at baseline and at the end of the 12-week training. During this course of research, subjects are strongly advised to stay with their present lifestyle and medication.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 55 and 80 years with a confirmed diagnosis of type 2 diabetes mellitus (T2DM) and an HbA1c of ≥ 6.5% and ≤ 11%.

Exclusion Criteria:

* Individuals will be excluded if they have a history of any of the following conditions: cardiac arrest, complex dysrhythmias at rest, complicated myocardial infarction or revascularization procedure, presence of congestive failure, presence of angina, signs or symptoms of post-event myocardial ischemia, renal impairment or proteinuria, hepatic impairment, severe gout or hyperuricemia or uncontrolled hypertension, a fall within the last year, musculoskeletal impairment such as inability to walk independently (after stroke or serious arthritis), neurocognitive disorder, or other diseases that limit their ability to engage in physical activities will be excluded. Individuals enrolled in other physical training programs will also be excluded to ensure any true effect of the proposed intervention can be captured.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1C) | Baseline
  HbA1c can be used to evaluate how well-controlled blood sugar has been throughout exercise program. Blood tests will be performed by a nurse at the community center and HbA1c tests will be conducted by a private medical laboratory.
Glycated Hemoglobin (HbA1C) | 6 weeks
  HbA1c can be used to evaluate how well-controlled blood sugar has been throughout
Glycated Hemoglobin (HbA1C) | 12 weeks
  HbA1c can be used to evaluate how well-controlled blood sugar has been throughout

SECONDARY OUTCOMES:
Chair Stand Test | Baseline
  Testing lower body strength
Chair Stand Test | 6 weeks
  Testing lower body strength
Chair Stand Test | 12 weeks
  Testing lower body strength
Arm Curl Test | Baseline
  Testing upper body strength
Arm Curl Test | 6 weeks
  Testing upper body strength
Arm Curl Test | 12 weeks
  Testing upper body strength
Chair Sit and Reach Test | Baseline
  Testing lower body flexibility
Chair Sit and Reach Test | 6 weeks
  Testing lower body flexibility
Chair Sit and Reach Test | 12 weeks
  Testing lower body flexibility
Back Scratch Test | Baseline
  Testing upper body flexibility
Back Scratch Test | 6 weeks
  Testing upper body flexibility
Back Scratch Test | 12 weeks
  Testing upper body flexibility
8-Foot Up and Go Test | Baseline
  Testing agility
8-Foot Up and Go Test | 6 weeks
  Testing agility
8-Foot Up and Go Test | 12 weeks
  Testing agility
Quadriceps strength | Baseline
  A handheld dynamometer will be used to assess quadriceps strength.
Quadriceps strength | 6 weeks
  A handheld dynamometer will be used to assess quadriceps strength.
Quadriceps strength | 12 weeks
  A handheld dynamometer will be used to assess quadriceps strength.
Hamstring Strength. | Baseline
  A handheld dynamometer will be used to assess hamstring strength.
Hamstring Strength. | 6 weeks
  A handheld dynamometer will be used to assess hamstring strength.
Hamstring Strength. | 12 weeks
  A handheld dynamometer will be used to assess hamstring strength.
Aerobic Capacity | Baseline
  The six-minute walk test will be conducted to assess aerobic capacity.
Aerobic Capacity | 6 weeks
  The six-minute walk test will be conducted to assess aerobic capacity.
Aerobic Capacity | 12 weeks
  The six-minute walk test will be conducted to assess aerobic capacity.
Exercise Compliance | Baseline
  Participant's compliance to the training program will be measured using Quartrics, a web-based survey system. Participants will receive a verbal reminder from research assistants to attend training sessions.
Exercise Compliance | 6 weeks
  Participant's compliance to the training program will be measured using Quartrics, a web-based survey system. Participants will receive a verbal reminder from research assistants to attend training sessions.
Exercise Compliance | 12 weeks
  Participant's compliance to the training program will be measured using Quartrics, a web-based survey system. Participants will receive a verbal reminder from research assistants to attend training sessions.
Balance | Baseline
  The Mini Balance Evaluation Systems Test (Mini-BEST) will be used to assess participant's ability to safely balance during a series of predetermined tasks.
Balance | 6 weeks
  The Mini Balance Evaluation Systems Test (Mini-BEST) will be used to assess participant's ability to safely balance during a series of predetermined tasks.
Balance | 12 weeks
  The Mini Balance Evaluation Systems Test (Mini-BEST) will be used to assess participant's ability to safely balance during a series of predetermined tasks.
Postural sway | Baseline
  Postural sway will be evaluated using a force plate, which is an instrument to measure static balance and dynamic balance. Postural sway will be assessed under both eyes opened and closed conditions.
Postural sway | 6 weeks
  Postural sway will be evaluated using a force plate, which is an instrument to measure static balance and dynamic balance. Postural sway will be assessed under both eyes opened and closed conditions.
Postural sway | 12 weeks
  Postural sway will be evaluated using a force plate, which is an instrument to measure static balance and dynamic balance. Postural sway will be assessed under both eyes opened and closed conditions.
Forward Version of Digit-Span Test | Baseline
  Forward Version of Digit-Span Test will be used to assess short-term memory. Score ranges from 0 to 14. The higher score indicates the better memory.
Forward Version of Digit-Span Test | 6 weeks
  Forward Version of Digit-Span Test will be used to assess short-term memory. Score ranges from 0 to 14. The higher score indicates the better memory.
Forward Version of Digit-Span Test | 12 weeks
  Forward Version of Digit-Span Test will be used to assess short-term memory. Score ranges from 0 to 14. The higher score indicates the better memory.
Backward Version of Digit-Span Test | Baseline
  Backward Version of Digit-Span Test will be used to assess short-term memory. Score ranges from 0 to 14. The higher score indicates the better memory.
Backward Version of Digit-Span Test | 6 weeks
  Backward Version of Digit-Span Test will be used to assess short-term memory. Score ranges from 0 to 14. The higher score indicates the better memory.
Backward Version of Digit-Span Test | 12 weeks
  Backward Version of Digit-Span Test will be used to assess short-term memory. Score ranges from 0 to 14. The higher score indicates the better memory.
Executive Function | Baseline
  Wechsler Adult Intelligence Scale Digit-Symbol-Coding will be used to assess the executive function. The score ranges from 0 to 133. The higher score indicate the better executive function.
Executive Function | 6 weeks
  Wechsler Adult Intelligence Scale Digit-Symbol-Coding will be used to assess the executive function. The score ranges from 0 to 133. The higher score indicate the better executive function.
Executive Function | 12 weeks
  Wechsler Adult Intelligence Scale Digit-Symbol-Coding will be used to assess the executive function. The score ranges from 0 to 133. The higher score indicate the better executive function.
Depression | Baseline
  The 17-item version of the English and Chinese Diabetes Distress Scale will be used to assess the mental health status. The mean item score ranges from 1 to 6. The mean item score of 3 or above (moderate distress) is considered as the level of distress worthy of clinical attention.
Depression | 6 weeks
  The 17-item version of the English and Chinese Diabetes Distress Scale will be used to assess the mental health status. The mean item score ranges from 1 to 6. The mean item score of 3 or above (moderate distress) is considered as the level of distress worthy of clinical attention.
Depression | 12 weeks
  The 17-item version of the English and Chinese Diabetes Distress Scale will be used to assess the mental health status. The mean item score ranges from 1 to 6. The mean item score of 3 or above (moderate distress) is considered as the level of distress worthy of clinical attention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request.